CLINICAL TRIAL: NCT06585956
Title: The Role of Physician-Patient Communication Through Mobile Phone Application in Preventing Emergency Room Admissions After Circumcision: a Randomized Prospective Study
Brief Title: Prevent Post-discharge Hospital Admissions Using Mobile Phone App
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University Hospital (Other)
Responsible Party: Principal Investigator, İsmail Emre ERGİN, Phd, Cumhuriyet University Hospital
Other Study IDs: SCU-UR-IEE-06
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Surgery
Keywords: Anxiety; Patient Readmission; Circumcission; Telemedicine
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Communication Group: Physician-Patient Communication Group
  Interventions: Behavioral: Comminication via Telemedicine
- Non-Communication Group: Physician-Patient Non-Communication Group
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Comminication via Telemedicine — Comminication via Telemedicine With Patients
  Groups: Communication Group
Behavioral: Information — Informing the patient and their relatives
  Groups: Non-Communication Group

SUMMARY:
The investigators aimed to assess the impact of a mobile phone application facilitating real-time visual and verbal communication on reducing emergency room admissions following circumcision.

DETAILED DESCRIPTION:
Today, communication devices make our lives easier and provide convenience in the healthcare sector. Some studies have mentioned that a definitive diagnosis can be made with digital photographs and video images in children with normal findings at the time of examination, and further diagnostic tests become unnecessary . Readmission to the hospital after surgery, especially in children, is a situation that increases the level of anxiety. The use of smart device applications to evaluate both the operation site and functional results after many surgical procedures has reduced the number of re-applications and anxiety levels of patients . Through communication, the patient can articulate their needs to the physician, either verbally or visually, and with the assistance of the physician, navigate through this process much more smoothly. In our randomized prospective study, the investigators aimed to assess the role of a mobile phone application facilitating real-time visual and verbal communication, as well as instant information exchange, in reducing emergency room and urology policlinic admissions due to potential complications after circumcision.

ELIGIBILITY:
Inclusion Criteria:

* Circumcision

Exclusion Criteria:

* hypospadias
* cryptoorchidism
* bleeding diathesis

Ages: 1 Year to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male
Study Population: Cases of circumcision
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The Role of Physician-Patient Communication through Mobile Phone Application in Preventing Emergency Room Admissions after Circumcision: A Randomized Prospective Study | To estimate the change in the readmission rate during the participants; recovery period (2 months)
  Predicting reduction in patient readmission rate using telemedicine assistance

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet Univercity, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No